CLINICAL TRIAL: NCT00852969
Title: Does Raising HDL-C With Niacin Improve Endothelial Function in Early CKD?
Brief Title: Niacin and Endothelial Function in Early CKD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 5R21DK077368 (NIH); 5R21DK077368-02 (NIH)
Record Dates: First submitted 2009-02-26; First posted 2009-02-27 (Estimated); Results first posted 2014-05-06 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2014-04

CONDITIONS: Chronic Kidney Disease
Keywords: Chronic Kidney Disease; Niacin; HDL; Endothelial Function
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Niacin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Niacin (Active Comparator)
  Interventions: Drug: Niacin
- Placebo (Placebo Comparator)
  Interventions: Drug: Active Placebo

INTERVENTIONS:
Drug: Niacin — 1000 mg tablets once per day
  Other Names: Niaspan
  Arms: Niacin
Drug: Active Placebo — 100 mg Niacin tablets once per day
  Arms: Placebo

SUMMARY:
The purpose of this study is to obtain information on whether raising levels of HDL-cholesterol (the "good" cholesterol) can improve how blood vessels work in kidney disease. This may help us understand the causes leading to high rates of heart disease in kidney disease and also ways to reduce this risk.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CKD Stage 2 (GFR >60 and microalbuminuria/proteinuria) and Stage 3-4 (GFR 15-30)
* HDL-cholesterol <50 for men and <55 for women
* If taking a statin, stable dose for past one month
* Glucose <200 mg/dL and HbA1c <9%
* Transplant recipients who are in stage 2-3 CKD; 1-year post transplant; and have had no rejection episodes in the 6-months prior to study entry

Exclusion Criteria:

* Hospitalization within prior 3 months
* Any of the following conditions:

  * uncontrolled peptic ulcer disease
  * active liver disease OR abnormal SGOT/SGPT
  * history of adverse reaction to niacin
  * contra-indication to aspirin
  * concurrent fibrate therapy
  * history of gout
  * serum phosphorus levels below 2.7mg/dl
* Nursing
* Pregnancy

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-08; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Sarnak, MD, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients were recruited at Tufts Medical Center. Dates of recruitment were 9/2008 to 11/2011
Pre-assignment Details: There was no washout period. Patients receiving Niacin were excluded from the study.
Groups:
- Niacin: Niacin : 1000 mg tablets once per day
- Placebo: Active Placebo : 100 mg Niacin tablets once per day. Placebo tablets had same appearance
Period: Overall Study
Arm/Group | Niacin | Placebo
Started | 15 | 15
Completed | 15 | 13
Not Completed | 0 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: These were the number of individuals who agreed to be randomized for the study
Groups:
- Total: Total of all reporting groups
Arm/Group | Niacin | Placebo | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 13 | 23
  >=65 years | 5 | 2 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.1 (10.9) | 50.4 (11.9) | 54.2 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 11 | 17
  Male | 9 | 4 | 13
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Change in the Flow Mediated Dilation From Baseline
Description: Flow mediated dilation by brachial artery reactivity at baseline versus 14 weeks
Time Frame: 14 weeks since baseline
Measure: Mean (95% Confidence Interval); unit: absolute percent change
Arm/Group | Niacin | Placebo
Number analyzed (Participants) | 15 | 13
absolute percent change | 3.07 [-2.36 to 8.50] | 1.37 [-6.81 to 9.56]
Statistical Analysis 1: Comparison: Niacin vs Placebo; Test type: Superiority or Other; p = 0.71, t-test, 2 sided; Mean Difference (Net) = -1.69, 95% CI 2-sided [-10.79 to 7.41]

2. Secondary Outcome: Change in HDL-C From Baseline to 14 Weeks
Time Frame: 14 weeks since baseline
Measure: Mean (95% Confidence Interval); unit: mg/dl
Arm/Group | Niacin | Placebo
Number analyzed (Participants) | 15 | 15
mg/dl | 5.22 [1.19 to 9.25] | 2.74 [-0.13 to 5.61]
Statistical Analysis 1: Comparison: Niacin vs Placebo; Test type: Superiority or Other; p = 0.29, t-test, 2 sided; Mean Difference (Net) = -2.48, 95% CI 2-sided [-7.20 to 2.24]

ADVERSE EVENTS:
Time Frame: During the trial up to 14 weeks
Arm/Group | Niacin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 10/15 | 5/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Niacin (N=15) | Placebo (N=15)
flushing (Skin and subcutaneous tissue disorders) | 10 (10) | 5 (5)
diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
constipation (Gastrointestinal disorders) | 0 (0) | 5 (5)
nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
joint pains (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No